CLINICAL TRIAL: NCT04878822
Title: Prospective, Cohort, Non-interventional, Single-center Clinical Study of Immune Response Status to SARS-CoV-2 / Covid-19 Vaccination in Patients With Haematological Malignancies.
Brief Title: Immunogenicity of Covid-19 Vaccination for Patients With Hematological Malignancies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Francesco Passamonti, Principal Investigator, Ospedale di Circolo - Fondazione Macchi
Other Study IDs: ImmunoHaema-COVID-VAX-21
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-05

CONDITIONS: Immunogenicity; Hematological Malignancies; Covid-19; Vaccine Response Impaired
Keywords: Hematological Malignancies; Covid-19; SARS-CoV-2; Comirnaty; Moderna; Vaxzevria; Janssen; Efficacy vaccination
MeSH Terms: conditions — Hematologic Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Covid-19 is associated with a mortality rate of 33-37% in patients with hematological malignancies.

At present, the anti-SARS-CoV-2 vaccination represents the most effective strategy for the prevention of Covid-19. Patients with malignancies were excluded from the trials leading to the approval of Comirnaty, Moderna, Vaxzevria and Janssen vaccines. The immunogenicity of these vaccines in immunocompromised patients or with hematological malignancies is an unmet clinical need.

The aim of the study is to evaluate the efficacy of vaccination in adult patients with hematological malignancies, who received vaccination according to Italian rules and were in treatment at the Hematology Unit of Varese, Italy Efficacy will be evaluated in terms of serological response, cellular-mediated immune response and prevention of Covid-19.

The duration of the study will be 24 months.

DETAILED DESCRIPTION:
Covid-19 is associated with a mortality rate of 33-37% in patients with hematological malignancies (Passamonti et al, 2020; Garcia-Suarez et al, 2020). Currently, there is little information on the serological response following SARS-Cov-2 infection in this specific population.

At present, the anti-SARS-CoV-2 vaccination represents the most effective strategy for the prevention of Covid-19. The anti-SARS-CoV-2 vaccines currently approved by the European Medicines Agency (EMA) and the Italian Medicines Agency (Agenzia Italiana del Farmaco, AIFA) are: the BNT162b2 SARS-Cov-2 (Pfizer-BioNTech, Comirnaty) vaccine, the mRNA-1273 SARS-Cov-2 (Moderna) vaccine, the ChAdOx1 nCoV-19 (Vaxzevria) vaccine, and the Ad26.COV2.S (Janssen) vaccine.

The double-dose regimen of Pfizer-BioNTech vaccine showed 95% efficacy at preventing Covid-19 (Polack et al, 2020), the double-dose regimen of Moderna vaccine showed 94.1% efficacy (Baden et al, 2021), the double-dose regimen of Vaxzevria vaccine showed 70.4% efficacy (Voysey et al, 2021), while the single-dose regimen of Janssen vaccine was found to be 66.1% effective (Sadoff et al, 2021).

The Italian national Covid-19 vaccination plan included patients with active malignancies in the second priority group, recognizing the importance of protecting this vulnerable population from SARS-Cov-2 infection. Since vaccine clinical trials excluded patients with malignancies and patients undergoing immunosuppressive therapies, the immunological response to anti-SARS-CoV-2 vaccines in these patients is currently unknown.

In this prospective, cohort, non-interventional study, our objective is to evaluate both the humoral and the cellular immune response to anti-SARS-CoV-2 vaccination in adults with hematological malignancies. For each patient the immune response will be evaluated after a minimum of 28 days from the completion of the vaccination regimen. Then, it will be reassessed after 6 and 12 months. In our center, the humoral immune response will be assessed by using the DiaSorin's LIAISON SARS-CoV-2 S1/S2 IgG test, which quantifies the level of anti-SARS-CoV-2 IgG antibodies that are active against the S1 and S2 subunits of the S protein. The cell-mediated immune response will be assessed on peripheral blood cells through a phenotypic and functional analysis by flow cytometry and through the ELISPOT test. Each patients will sign an informed consensus for the participation. The total duration of the study will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* History of hematological neoplasia (myeloid neoplasms, lymphoid neoplasms, plasma cell dyscrasias).
* Active hematological neoplasm.

Exclusion Criteria:

* Hematological diseases, other than hematological malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with hematological malignancies who have received the anti-SARS-CoV2 / Covid-19 vaccination, with or without previous Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the humoral immune response to SARS-CoV-2 / Covid-19 vaccination. | 1 month after completion of vaccination
  The percentage of patients with positive antibody titer (≥ 12 AU / mL) after at least 28 days from vaccination.

SECONDARY OUTCOMES:
To evaluate the humoral immune response to SARS-CoV-2 / Covid-19 vaccination according to the disease and its status. | 1 month after completion of vaccination
  The percentage of patients with positive antibody titer (≥ 12 AU / mL) after at least 28 days from vaccination in myeloid, lymphoid and plasma cell dyscrasias sub-categorized by status of disease, status and type of treatment.
To evaluate the humoral immune response to SARS-CoV-2 / Covid-19 vaccination according to the type of vaccination. | 1 month after completion of vaccination
  The percentage of patients with positive antibody titer (≥ 12 AU / mL) after at least 28 days from vaccination described by vaccine brand (currently Comirnaty, Moderna, Vaxzevria, Janssen).
To assess the antibody titer at least 28 days after the SARS-CoV-2 / Covid-19 vaccination. | 1 month after completion of vaccination
  The distribution and median of the antibody titer at least 28 days after vaccination.
To evaluate the persistence of the antibody titer after vaccination. | 28 days, 6 and 12 months after completion of vaccination
  The difference between the antibody titer at 28 days and at 6 and 12 months after vaccination.
To evaluate the cellular immune response to SARS-CoV-2 / Covid-19 vaccination. | 28 days, 6 and 12 months after completion of vaccination
  The percentage of patients who generated immune cells with IFN-gamma cytokine response after at least 28 days, 6 and 12 months after vaccination.
To evaluate the clinical efficacy of the anti SARS-CoV-2 / Covid-19 vaccination. | 28 days, 6 and 12 months after completion of vaccination
  The percentage of patients with any among: 1) positive molecular swab by RT-PCR, 2) documented symptomatic Covid-19 disease; 3) hospitalization for Covid-19; 4) documented severe Covid-19 disease; 5) death from Covid-19 despite vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Passamonti, MD, Principal Investigator — Ospedale di Circolo e Fondazione Macchi, ASST Sette Laghi, Varese, Italy
Locations (1):
- UOC Ematologia, ASST Sette Laghi, Osp. Di Circolo e Fondazione Macchi, Varese, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Passamonti F, Cattaneo C, Arcaini L, Bruna R, Cavo M, Merli F, Angelucci E, Krampera M, Cairoli R, Della Porta MG, Fracchiolla N, Ladetto M, Gambacorti Passerini C, Salvini M, Marchetti M, Lemoli R, Molteni A, Busca A, Cuneo A, Romano A, Giuliani N, Galimberti S, Corso A, Morotti A, Falini B, Billio A, Gherlinzoni F, Visani G, Tisi MC, Tafuri A, Tosi P, Lanza F, Massaia M, Turrini M, Ferrara F, Gurrieri C, Vallisa D, Martelli M, Derenzini E, Guarini A, Conconi A, Cuccaro A, Cudillo L, Russo D, Ciambelli F, Scattolin AM, Luppi M, Selleri C, Ortu La Barbera E, Ferrandina C, Di Renzo N, Olivieri A, Bocchia M, Gentile M, Marchesi F, Musto P, Federici AB, Candoni A, Venditti A, Fava C, Pinto A, Galieni P, Rigacci L, Armiento D, Pane F, Oberti M, Zappasodi P, Visco C, Franchi M, Grossi PA, Bertu L, Corrao G, Pagano L, Corradini P; ITA-HEMA-COV Investigators. Clinical characteristics and risk factors associated with COVID-19 severity in patients with haematological malignancies in Italy: a retrospective, multicentre, cohort study. Lancet Haematol. 2020 Oct;7(10):e737-e745. doi: 10.1016/S2352-3026(20)30251-9. Epub 2020 Aug 13. PMID 32798473
- [Background] Garcia-Suarez J, de la Cruz J, Cedillo A, Llamas P, Duarte R, Jimenez-Yuste V, Hernandez-Rivas JA, Gil-Manso R, Kwon M, Sanchez-Godoy P, Martinez-Barranco P, Colas-Lahuerta B, Herrera P, Benito-Parra L, Alegre A, Velasco A, Matilla A, Alaez-Uson MC, Martos-Martinez R, Martinez-Chamorro C, Susana-Quiroz K, Del Campo JF, de la Fuente A, Herraez R, Pascual A, Gomez E, Perez-Oteyza J, Ruiz E, Alonso A, Gonzalez-Medina J, Martin-Buitrago LN, Canales M, Gonzalez-Gascon I, Vicente-Ayuso MC, Valenciano S, Roa MG, Monteliu PE, Lopez-Jimenez J, Escobar CE, Ortiz-Martin J, Diez-Martin JL, Martinez-Lopez J; Asociacion Madrilena de Hematologia y Hemoterapia (AMHH). Impact of hematologic malignancy and type of cancer therapy on COVID-19 severity and mortality: lessons from a large population-based registry study. J Hematol Oncol. 2020 Oct 8;13(1):133. doi: 10.1186/s13045-020-00970-7. PMID 33032660
- [Background] Roeker LE, Knorr DA, Pessin MS, Ramanathan LV, Thompson MC, Leslie LA, Zelenetz AD, Mato AR. Anti-SARS-CoV-2 antibody response in patients with chronic lymphocytic leukemia. Leukemia. 2020 Nov;34(11):3047-3049. doi: 10.1038/s41375-020-01030-2. Epub 2020 Aug 27. No abstract available. PMID 32855439
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Background] Boyarsky BJ, Werbel WA, Avery RK, Tobian AAR, Massie AB, Segev DL, Garonzik-Wang JM. Immunogenicity of a Single Dose of SARS-CoV-2 Messenger RNA Vaccine in Solid Organ Transplant Recipients. JAMA. 2021 May 4;325(17):1784-1786. doi: 10.1001/jama.2021.4385. PMID 33720292
- [Background] Sadoff J, Gray G, Vandebosch A, Cardenas V, Shukarev G, Grinsztejn B, Goepfert PA, Truyers C, Fennema H, Spiessens B, Offergeld K, Scheper G, Taylor KL, Robb ML, Treanor J, Barouch DH, Stoddard J, Ryser MF, Marovich MA, Neuzil KM, Corey L, Cauwenberghs N, Tanner T, Hardt K, Ruiz-Guinazu J, Le Gars M, Schuitemaker H, Van Hoof J, Struyf F, Douoguih M; ENSEMBLE Study Group. Safety and Efficacy of Single-Dose Ad26.COV2.S Vaccine against Covid-19. N Engl J Med. 2021 Jun 10;384(23):2187-2201. doi: 10.1056/NEJMoa2101544. Epub 2021 Apr 21. PMID 33882225
- See also: Description and mechanism of action of COVID-19 m-RNA vaccines authorised by EMA and AIFA — http://www.aifa.gov.it/vaccini-mrna
- See also: The latest updates on the COVID-19 pandemic from the European Medicines Agency (EMA) — http://www.ema.europa.eu/en/human-regulatory/overview/public-health-threats/coronavirus-disease-covid-19/covid-19-latest-updates
- See also: Italian plan for Sar-CoV-2 vaccination — https://www.trovanorme.salute.gov.it/norme/renderPdf.spring?seriegu=SG&datagu=24/03/2021&redaz=21A01802&artp=1&art=1&subart=1&subart1=10&vers=1&prog=002